CLINICAL TRIAL: NCT02848326
Title: A Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel-Group Study To Evaluate The Efficacy, Safety, And Tolerability Of Multiple Dosing Regimens Of Oral AGN-241689 In Episodic Migraine Prevention
Brief Title: Efficacy, Safety, and Tolerability of Multiple Dosing Regimens of Oral Atogepant (AGN-241689) in Episodic Migraine Prevention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CGP-MD-01
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo-matching atogepant capsule orally twice daily in the morning and in the evening for 12 weeks.
  Interventions: Drug: Placebo-matching Atogepant
- Atogepant 10 mg QD (Experimental): Atogepant 10 mg capsule orally once daily (QD) in the morning and one placebo-matching atogepant capsule orally once daily in the evening for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo-matching Atogepant
- Atogepant 30 mg QD (Experimental): Atogepant 30 mg capsule orally once daily in the morning and one placebo-matching atogepant capsule orally once daily in the evening for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo-matching Atogepant
- Atogepant 30 mg BID (Experimental): Atogepant 30 mg capsule orally twice daily (BID); 1 capsule in the morning and 1 capsule in the evening for 12 weeks.
  Interventions: Drug: Atogepant
- Atogepant 60 mg QD (Experimental): Atogepant 60 mg capsule orally once daily in the morning and one placebo-matching atogepant capsule orally in the evening for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo-matching Atogepant
- Atogepant 60 mg BID (Experimental): Atogepant 60 mg capsule orally twice daily; 1 capsule in the morning and 1 capsule in the evening for 12 weeks.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Atogepant capsule.
  Other Names: AGN-241689
  Arms: Atogepant 10 mg QD; Atogepant 30 mg BID; Atogepant 30 mg QD; Atogepant 60 mg BID; Atogepant 60 mg QD
Drug: Placebo-matching Atogepant — Placebo-matching atogepant capsule.
  Arms: Atogepant 10 mg QD; Atogepant 30 mg QD; Atogepant 60 mg QD; Placebo

SUMMARY:
This study will evaluate the safety and tolerability of the following doses of atogepant (AGN-241689): 10 mg once daily (QD), 30 mg QD, 30 mg twice daily (BID), 60 mg QD, and 60 mg BID for the prevention of episodic migraine and will characterize the dose/response relationship.

ELIGIBILITY:
Inclusion Criteria:

* Has at least a 1-year history of migraine with or without aura
* Age of the patient at the time of migraine onset < 50 years
* History of 4 to 14 migraine days (migraine/probable migraine headache days) per month on average in the 3 months prior to Visit 1 in the Investigator's judgment
* Demonstrated compliance with e-diary

Exclusion Criteria:

* Has a history of migraine accompanied by diplopia or decreased level of consciousness and retinal migraine
* Has a current diagnosis of chronic migraine, new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy
* Difficulty distinguishing migraine headache from other headaches
* Has a history of malignancy in the prior 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Has a history of gastric or small intestinal surgery, or has a disease that causes malabsorption
* Has a history of hepatitis within previous 6 months
* Usage of opioids or barbiturates > 2 days/month, triptans or ergots ≥ 10 days/month, or simple analgesics (eg, aspirin, non-steroidal anti-inflammatory drugs [NSAIDs], acetaminophen) ≥ 15 days/month in the 3 months prior to Visit 1
* Pregnant or nursing females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Trugman, MD, Study Director — Allergan
Locations (75):
- United States (75):
  - Achieve Clinical Research, Birmingham, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - The Research Center of Southern California, LLC, Carlsbad, California
  - Neuro-Pain Medical Center, Inc, Fresno, California
  - Irvine Center for Clinical Research, Irvine, California
  - Downtown LA Research Center, Inc., Los Angeles, California
  - Excell Research, Oceanside, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Diablo Clinical Research Inc, Walnut Creek, California
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Hartford Headache Center, East Hartford, Connecticut
  - Associated Neurologists of Southern Connecticut, P. C., Fairfield, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - The George Washington University, Washington D.C., District of Columbia
  - Clinical Research South Florida, Coral Gables, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Suncoast Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Palm Beach Neurological Center / Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Infinity Clinical Research LLC, Sunrise, Florida
  - Meridien Research, Tampa, Florida
  - Neurology Research Institute Palm Beach, West Palm Beach, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Radiant Research, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Pediatric and Adolescent NeuroDevelopmental Associates (PANDA) Neurology, Sandy Springs, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Healthcare Research Network II, LLC, Blue Island, Illinois
  - Rowe Neurology Institute, Lenexa, Kansas
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Medvadis Research Corporation, Watertown, Massachusetts
  - New England Regional Headache Center, Worcester, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Mercy Research, Springfield, Missouri
  - Clinvest, Springfield, Missouri
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Altea Research Institute, Las Vegas, Nevada
  - Renown Institute for Neuroscience, Reno, Nevada
  - Hassman Research Institute - NJ, Berlin, New Jersey
  - Amici Clinical Research, Warren Township, New Jersey
  - DENT Neurosciences Research Center, Amherst, New York
  - Radiant Research, Inc., Jamaica, New York
  - Carolina Headache Institute, Durham, North Carolina
  - Wake Research Associates LLC, Raleigh, North Carolina
  - Ohio Clinical Research, LLC, Willoughby Hills, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Cns Healthcare, Memphis, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Tekton Research, Austin, Texas
  - DermResearch Inc, Austin, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - Synexus US, L.P. Formally known as Texas Pharmaceutical Research, LP, DBA Research Across America, Dallas, Texas
  - Central Texas Neurology Consultant, Round Rock, Texas
  - Radiant Research, San Antonio Center for Clinical Research, San Antonio, Texas
  - Road Runner Research LTD, San Antonio, Texas
  - ClinPoint Trials, LLC, Waxahachie, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Women's Clinical Research Center, Seattle, Washington
  - Kingfisher Cooperative, LLC, Spokane, Washington

REFERENCES:
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Peterlin BL, Bond DS, Ailani J, Dodick DW, Liu Y, De Abreu Ferreira R, Smith JH, Dabruzzo B, Goadsby PJ, Trugman JM. Weight loss with atogepant during the preventive treatment of migraine: A pooled analysis. Cephalalgia. 2024 Dec;44(12):3331024241299753. doi: 10.1177/03331024241299753. PMID 39648629
- [Derived] Rizzoli P, Marmura MJ, Robblee J, McVige J, Sacco S, Nahas SJ, Ailani J, De Abreu Ferreira R, Ma J, Smith JH, Dabruzzo B, Ashina M. Safety and tolerability of atogepant for the preventive treatment of migraine: a post hoc analysis of pooled data from four clinical trials. J Headache Pain. 2024 Mar 11;25(1):35. doi: 10.1186/s10194-024-01736-z. PMID 38462625
- [Derived] Goadsby PJ, Dodick DW, Ailani J, Trugman JM, Finnegan M, Lu K, Szegedi A. Safety, tolerability, and efficacy of orally administered atogepant for the prevention of episodic migraine in adults: a double-blind, randomised phase 2b/3 trial. Lancet Neurol. 2020 Sep;19(9):727-737. doi: 10.1016/S1474-4422(20)30234-9. PMID 32822633
- See also: http://www.allerganclinicaltrials.com — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants diagnosed with migraine, with or without aura were enrolled in one of 6 treatment arms: placebo, or atogepant 10 mg once daily (QD), 30 mg QD, 60 mg QD, 30 mg twice daily (BID), or 60 mg BID.
Groups:
- Placebo: Placebo-matching atogepant capsules orally twice daily in the morning and in the evening for 12 weeks.
Period: Treatment Period
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
Started | 186 | 94 | 185 | 187 | 89 | 93
Safety Population: Received Study Drug | 186 | 93 | 183 | 186 | 86 | 91
Completed | 148 | 80 | 149 | 164 | 70 | 73
Not Completed | 38 | 14 | 36 | 23 | 19 | 20
Not completed — Adverse Event | 5 | 4 | 11 | 6 | 5 | 7
Not completed — Withdrawal of Consent | 20 | 6 | 9 | 6 | 9 | 6
Not completed — Lost to Follow-up | 5 | 1 | 11 | 7 | 2 | 3
Not completed — Pregnancy | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 4 | 3 | 4 | 2 | 3 | 3
Not completed — Non-compliance with Study Drug | 4 | 0 | 0 | 1 | 0 | 0
Period: Safety Follow-up Period
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
Started | 161 | 84 | 156 | 169 | 77 | 82
Completed | 157 | 83 | 153 | 169 | 76 | 77
Not Completed | 4 | 1 | 3 | 0 | 1 | 5
Not completed — Withdrawal of Consent | 0 | 1 | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 4 | 0 | 2 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID | Total
Number analyzed (Participants) | 186 | 93 | 183 | 186 | 86 | 91 | 825
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (11.7) | 39.4 (12.4) | 41.0 (13.6) | 40.4 (11.7) | 38.5 (11.2) | 39.7 (11.9) | 40.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 82 | 166 | 156 | 73 | 83 | 714
  Male | 32 | 11 | 17 | 30 | 13 | 8 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 137 | 69 | 145 | 133 | 73 | 71 | 628
  Black or African American | 45 | 20 | 29 | 44 | 11 | 19 | 168
  Asian | 1 | 1 | 2 | 3 | 1 | 0 | 8
  American Indian or Alaska Native | 3 | 0 | 1 | 2 | 0 | 0 | 6
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Multiple Races | 0 | 3 | 4 | 4 | 1 | 1 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 15 | 32 | 25 | 13 | 13 | 127
  Not Hispanic or Latino | 157 | 78 | 151 | 161 | 73 | 78 | 698
Migraine Days (Migraine/Probable Migraine Headache Days) [Mean (Standard Deviation); unit: migraine days per month] — A migraine day was any calendar day on which the participant experienced a migraine headache qualified by duration and acute symptomatic medication use. The 4-week migraine days=total number of reported migraine days in diary divided by total number of days with diary records in each 4-week period multiplied by 28. Population: Modified-intent-to-treatment (mITT) Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of diary data, and had at least 1 evaluable post-baseline 4-week (Weeks 1-4, 5-8, and 9-12) of diary data.
  migraine days per month
    number analyzed (Participants) | 178 | 92 | 182 | 177 | 79 | 87 | 795
    (all) | 7.81 (2.51) | 7.63 (2.51) | 7.64 (2.37) | 7.74 (2.59) | 7.38 (2.43) | 7.62 (2.56) | 7.67 (2.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days (Migraine/Probable Migraine Headache Days) Across the 12-Week Treatment Period
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache qualified by duration and acute symptomatic medication use. The 4-week migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4- week period and multiplied by 28. Each 4-week period was averaged. Negative change from Baseline indicates improvement.
Time Frame: Baseline (First 28 Days of Screening/Baseline Period) to Week 12
Population: MITT Population included all randomized participants who received at least 1 dose of study treatment, had an evaluable baseline period of diary data, and had at least 1 evaluable post-baseline 4-week (Weeks 1-4, 5-8, and 9-12) of diary data.
Measure: Least Squares Mean (Standard Error); unit: migraine days per month
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
Number analyzed (Participants) | 178 | 92 | 182 | 177 | 79 | 87
migraine days per month | -2.85 (0.23) | -4.00 (0.32) | -3.76 (0.23) | -3.55 (0.23) | -4.23 (0.35) | -4.14 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg QD; Test type: Superiority; p = 0.0039, MMRM — Mixed-effects model for repeated measures (MMRM) model included baseline monthly migraine days as a covariate, treatment group and visit (month) as fixed factors, and treatment group-by-visit and baseline-by-visit as interaction terms; Least squares mean difference = -1.15, 95% CI 2-sided [-1.93 to -0.37], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg QD; Test type: Superiority; p = 0.0056, MMRM — MMRM model included baseline monthly migraine days as a covariate, treatment group and visit (month) as fixed factors, and treatment group-by-visit and baseline-by-visit as interaction terms; Least squares mean difference = -0.91, 95% CI 2-sided [-1.55 to -0.27], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0325, MMRM — [p-value comment as in outcome 1, analysis 2]; Least squares mean difference = -0.70, 95% CI 2-sided [-1.35 to -0.06], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 1, analysis 2]; Least squares mean difference = -1.39, 95% CI 2-sided [-2.21 to -0.56], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: Placebo vs Atogepant 60 mg BID; Test type: Superiority; p = 0.0016, MMRM — [p-value comment as in outcome 1, analysis 2]; Least squares mean difference = -1.29, 95% CI 2-sided [-2.09 to -0.49], Standard Error of Mean 0.41

2. Secondary Outcome: Change From Baseline in Mean Monthly Headache Days Across the 12-Week Treatment Period
Description: Participants recorded daily total duration of a headache in a diary. A headache day is any calendar day on which the participant experienced a headache qualified by duration and acute symptomatic medication use. The 4-week (monthly) headache days was defined as the total number of reported headache days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Negative change from Baseline indicates improvement.
Time Frame: Baseline (First 28 Days of Screening/Baseline Period) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: headache days per month
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
Number analyzed (Participants) | 178 | 92 | 182 | 177 | 79 | 87
headache days per month | -2.93 (0.25) | -4.31 (0.35) | -4.17 (0.25) | -3.86 (0.25) | -4.23 (0.38) | -4.32 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg QD; Test type: Superiority; p = 0.0014, MMRM — MMRM model included baseline monthly headache days as a covariate, treatment group and visit (month) as fixed factors, and treatment group-by-visit and baseline-by-visit as interaction terms; Least squares mean difference = -1.38, 95% CI 2-sided [-2.23 to -0.54], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg QD; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 2, analysis 1]; Least squares mean difference = -1.24, 95% CI 2-sided [-1.94 to -0.55], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0087, MMRM — [p-value comment as in outcome 2, analysis 1]; Least squares mean difference = -0.94, 95% CI 2-sided [-1.64 to -0.24], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0044, MMRM — [p-value comment as in outcome 2, analysis 1]; Least squares mean difference = -1.30, 95% CI 2-sided [-2.20 to -0.41], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: Placebo vs Atogepant 60 mg BID; Test type: Superiority; p = 0.0017, MMRM — [p-value comment as in outcome 2, analysis 1]; Least squares mean difference = -1.39, 95% CI 2-sided [-2.26 to -0.53], Standard Error of Mean 0.44

3. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in Mean Monthly Migraine Days (Migraine/Probable Migraine Headache Days) Across the 12-Week Treatment Period
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache qualified by duration and acute symptomatic medication use. The 4-week migraine days=total number of reported migraine days in diary divided by total number of days with diary records in each 4-week period multiplied by 28. Each 4-week period was averaged.
Time Frame: Baseline (First 28 Days of Screening/Baseline Period) to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
Number analyzed (Participants) | 178 | 92 | 182 | 177 | 79 | 87
percentage of participants | 40.4 | 57.6 | 53.3 | 52.0 | 58.2 | 62.1
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg QD; Test type: Superiority; p = 0.0617, GLMM for repeated measures — Generalized linear mixed model (GLMM) for repeated measures with fixed factors(treatment group,visit), covariates(baseline migraine days), interactions(treatment group;baseline migraine days by visit) with an unstructured covariance matrix; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.98 to 2.31]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg QD; Test type: Superiority; p = 0.0369, GLMM for repeated measures — GLMM for repeated measures with fixed factors (treatment group, visit), covariates (baseline migraine days), interactions (treatment group by visit; baseline migraine days by visit) with an unstructured covariance matrix; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.02 to 2.08]
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0512, GLMM for repeated measures — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.00 to 2.03]
Statistical Analysis 4: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0113, GLMM for repeated measures — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.15 to 2.91]
Statistical Analysis 5: Comparison: Placebo vs Atogepant 60 mg BID; Test type: Superiority; p = 0.0019, GLMM for repeated measure — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.30 to 3.18]

4. Secondary Outcome: Change From Baseline in Mean Monthly Acute Medication Use Days Across the 12-Week Treatment Period
Description: Participants recorded allowed medication(s) to treat an acute migraine in the daily diary. The 4-week (monthly) acute medication use days was defined as the total number of reported acute medication use days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. A negative change from Baseline indicates improvement.
Time Frame: Baseline (First 28 Days of Screening/Baseline Period) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: acute medication use days per month
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
Number analyzed (Participants) | 178 | 92 | 182 | 177 | 79 | 87
acute medication use days per month | -2.42 (0.21) | -3.71 (0.29) | -3.86 (0.20) | -3.53 (0.21) | -3.77 (0.31) | -3.64 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg QD; Test type: Superiority; p = 0.0002, MMRM — MMRM model included baseline monthly acute medication use days as a covariate, treatment group and visit (month) as fixed factors, and treatment group-by-visit and baseline-by-visit as interaction terms; Least squares mean difference = -1.30, 95% CI 2-sided [-1.99 to -0.60], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg QD; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; Least squares mean difference = -1.44, 95% CI 2-sided [-2.01 to -0.87], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; Least squares mean difference = -1.11, 95% CI 2-sided [-1.68 to -0.54], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 4, analysis 1]; Least squares mean difference = -1.35, 95% CI 2-sided [-2.08 to -0.62], Standard Error of Mean 0.37
Statistical Analysis 5: Comparison: Placebo vs Atogepant 60 mg BID; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 4, analysis 1]; Least squares mean difference = -1.22, 95% CI 2-sided [-1.93 to -0.52], Standard Error of Mean 0.36

ADVERSE EVENTS:
Time Frame: Up to Week 16
Description: Safety population, all randomized participants who received at least 1 dose of study treatment, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | Atogepant 10 mg QD | Atogepant 30 mg QD | Atogepant 60 mg QD | Atogepant 30 mg BID | Atogepant 60 mg BID
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/93 | 0/183 | 0/186 | 0/86 | 0/91
Serious Adverse Events (participants affected / at risk) | 2/186 | 1/93 | 2/183 | 2/186 | 0/86 | 0/91
Other Adverse Events (participants affected / at risk) | 36/186 | 17/93 | 47/183 | 52/186 | 21/86 | 26/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Atogepant 10 mg QD (N=93) | Atogepant 30 mg QD (N=183) | Atogepant 60 mg QD (N=186) | Atogepant 30 mg BID (N=86) | Atogepant 60 mg BID (N=91)
Ureteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Atogepant 10 mg QD (N=93) | Atogepant 30 mg QD (N=183) | Atogepant 60 mg QD (N=186) | Atogepant 30 mg BID (N=86) | Atogepant 60 mg BID (N=91)
Fatigue (General disorders) | 6 | 1 | 3 | 5 | 2 | 9
Nausea (Gastrointestinal disorders) | 9 | 5 | 13 | 21 | 7 | 9
Constipation (Gastrointestinal disorders) | 4 | 2 | 10 | 9 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 14 | 6 | 13 | 9 | 4 | 6
Nasopharyngitis (Infections and infestations) | 4 | 3 | 10 | 14 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 3 | 3 | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02848326/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02848326/SAP_001.pdf